CLINICAL TRIAL: NCT03498989
Title: Effect of Early Feeding of Breast Milk Versus Formula Milk on Health Status of Preterm
Brief Title: Effect of Early Feeding of Breast Milk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AATaha, Paediatric, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Effect of early feeding
Record Dates: First submitted 2018-03-21; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Neonatal SEPSIS; Weight Gain; Feeding Disorder Neonatal
MeSH Terms: conditions — Neonatal Sepsis; Weight Gain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preterm formula milk neoborn (Experimental): will be given preterm formula milk
  Interventions: Other: preterm formula milk
- exclusive breast milk (Experimental): will be given exclusive breast milk
  Interventions: Other: exclusive breast milk

INTERVENTIONS:
Other: preterm formula milk — A. complete blood picture
  B. C-reactive protein
  C. Serum electrolytes
  D. Plain x-ray and abdominal ultrasound.
  Arms: preterm formula milk neoborn
Other: exclusive breast milk — exclusive breast milk
  Arms: exclusive breast milk

SUMMARY:
Breast milk is an extremely complex and highly variable biofliud that has evolved to nourish infants and protect them from disease whilst their own immune system matures. The composition of human breast milk changes in response to many factors, matching the infants requirement according to its age and other characteristics.

DETAILED DESCRIPTION:
Breast milk is an extremely complex and highly variable biofliud that has evolved to nourish infants and protect them from disease whilst their own immune system matures. The composition of human breast milk changes in response to many factors, matching the infants requirement according to its age and other characteristics.

Therefore, the composition of breast milk is widely believed to be specifically tailored by each mother to precisely reflect the requirements of her infant.

Human milk is uniquely suited to the human infant, both in its nutritional composition and in the non-nutritive bioactive factors that promote survival and healthy development.

Breast milk contains over 400 different proteins which perform a variety of functions; providing nutrition, possessing antimicrobial and immunomodulatory activities, as well as stimulating the absorption of nutrients.

The immune system of preterm infants is immature, placing them at increased risk for serious immune-related complications.

Human milk provides a variety of immune protective and immune maturation factors that are beneficial to the preterm infants poorly developed immune system. The most studied immune components in human milk include antimicrobial proteins, maternal leukocytes, immunoglobulins, cytokines and chemokines, oligosaccharides, gangliosides, nucleotides, and long-chain polyunsaturated fatty acids. There is growing evidence that these components contribute to the lower incidence of immune-related conditions in the preterm infant. Therefore, provision of these components in human milk, donor milk, or formula may provide immunologic benefits.

The effects of breast milk and breastfeeding on neurodevelopment may be quite different in very preterm infants than in those born at full term. Nutritionally, breast milk is considered the optimal food for full term infants. But preterm infants require fortification to match third trimester nutrient accretion rates.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age <37 weeks.
2. Birth weight >1000 gm.

Exclusion Criteria:

1. Gestational age 37 weeks.
2. Birth weight < 1000 gm.
3. Newborns with congenital anomalies.
4. Newborns with suspected metabolic diseases.
5. Newborns on mechanical ventilators.
6. Newborns with suspected neonatal sepsis.

Ages: 1 Week to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-06-21 (Estimated); Primary Completion 2019-03-21 (Estimated); Study Completion 2020-02-21 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 1 year
  All newborn well examine regards weight
  1. Necrotizing enterocolitis.
  2. Neonatal Sepsis.
  3. Weight gain.
  4. Feeding tolerance
Number of participants with complete blood pictures | 1 year
  All newborn are examine

REFERENCES:
- [Background] Fujita M, Roth E, Lo YJ, Hurst C, Vollner J, Kendell A. In poor families, mothers' milk is richer for daughters than sons: a test of Trivers-Willard hypothesis in agropastoral settlements in Northern Kenya. Am J Phys Anthropol. 2012 Sep;149(1):52-9. doi: 10.1002/ajpa.22092. Epub 2012 May 24. PMID 22623326
- [Background] Molinari CE, Casadio YS, Hartmann BT, Livk A, Bringans S, Arthur PG, Hartmann PE. Proteome mapping of human skim milk proteins in term and preterm milk. J Proteome Res. 2012 Mar 2;11(3):1696-714. doi: 10.1021/pr2008797. Epub 2012 Feb 22. PMID 22309230